CLINICAL TRIAL: NCT06976684
Title: Application of Extended Reality (XR)-Assisted CT-Guided Localization of Pulmonary Nodules in Thoracoscopic Sublobar Resection.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202502149RINB
Record Dates: First submitted 2025-04-24; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-04

CONDITIONS: Lung Cancers; Metaverse; Virtual Surgical Simulation; Extended Reality (XR)
Keywords: Metaverse; virtual surgical simulation; Extended Reality (XR); Pulmonary Nodules; Digital Twin
MeSH Terms: conditions — Lung Neoplasms; Multiple Pulmonary Nodules

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Extended Reality (XR)-Assisted CT-Guided Localization (Experimental)
  Interventions: Procedure: Extended Reality (XR)-Assisted CT-Guided Localization

INTERVENTIONS:
Procedure: Extended Reality (XR)-Assisted CT-Guided Localization — This study plans to collect approximately 20 localization cases from multiple centers within our hospital. Initially, two sets of preoperative simulated CT scans (at end-inhalation and end-exhalation) will be performed in the CT suite to construct a usable model of the surgical posture and the lesion. Subsequently, in the hybrid operating room, a digital twin model will be applied to the patient using a metaverse platform. Guided by virtual localization lines, percutaneous injection of Patent Blue dye will be carried out at end-exhalation for accurate marking of the lesion. Immediately after the injection, intraoperative CT within the hybrid operating room will be used to verify the localization. If the accuracy is suboptimal (with a deviation greater than 2 cm), standard CT-guided Patent Blue dye localization will be performed as a supplementary measure to complete the localization and proceed with surgery.

SUMMARY:
Reality (XR)-Assisted CT-Guided Localization

DETAILED DESCRIPTION:
With the widespread use of computed tomography (CT), lung nodules detected through screening have become increasingly smaller. These small nodules are often hidden within the lung parenchyma, making them difficult to visualize or palpate during surgery. As a result, nodule localization techniques have become critically important and are heavily relied upon by thoracic surgeons. Currently, CT-guided localization is the standard approach; however, this requires patients to move between the CT suite, the ward, and the operating room, which is highly inconvenient.

An alternative is the use of a one-stop hybrid operating room, which integrates imaging and surgery in a single space, but this solution is costly. This study aims to enroll 20 patients in a pilot investigation of using extended reality (XR)-guided localization in video-assisted thoracoscopic surgery (VATS) for lung nodule resection. By leveraging current XR technologies, a digital twin model will be superimposed onto the patient's body. Our team-developed virtual localization technique will then be used to mark the tumor site with dye, enabling surgeons to precisely excise the tumor with minimal tissue removal.

If successful, this technology has the potential to replace traditional CT-guided or hybrid operating room localization, thereby reducing patient inconvenience and financial burden, and ultimately achieving a streamlined and cost-effective surgical workflow.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 80 who are scheduled to undergo lung nodule resection surgery.
* Patients with lung nodules smaller than 2 cm that require preoperative localization.
* Patients with lung nodules located in the outer one-third of the lung.

Exclusion Criteria:

* Patients younger than 18 or older than 80 years.
* Patients requiring lobectomy.
* Patients who have not provided written informed consent.
* Vulnerable populations.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The Accuracy of Extended Reality (XR)-Assisted CT-Guided Localization | Immediatedly after Extended Reality (XR)-Assisted CT-Guided Localization
  Procedures in this study will be conducted in a hybrid operating room featuring cone-beam CT. The accuracy of XR-assisted CT-guided localization will be assessed immediately post-localization by employing cone-beam CT to ascertain the needle tip position and measure the distance to the target tumor.

SECONDARY OUTCOMES:
Assessment of perioperative outcomes | The study assessment time frame from XR-assisted CT-guided localization to discharge is approximately 3 to 7 days.
  Perioperative outcomes, including but not limited to intraoperative blood loss, localization time, and operative time, will be measured.

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data (IPD) collected during this study will generally not be shared with other researchers, primarily due to patient privacy considerations. However, limited access to de-identified IPD may be considered in exceptional cases upon a reasonable request.